CLINICAL TRIAL: NCT03756428
Title: Effects on Plantar Support After Deep Dry Needling in Posterior Tibial Muscle: Baropodometric Study
Brief Title: Effects on Plantar Support After Deep Dry Needling in Posterior Tibial Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, SERGIO MONTERO NAVARRO, Principal Investigator, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEU UCH 210
Record Dates: First submitted 2018-11-21; First posted 2018-11-28 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Movement Disorders
MeSH Terms: conditions — Movement Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep dry needling in tibialis posterior (Experimental): Deep dry needling will be applied in the tibialis posterior myofascial trigger point
  Interventions: Procedure: Deep dry needling in tibialis posterior
- Sham technique in tibialis posterior (Placebo Comparator): Placebo tibialis dry needling
  Interventions: Procedure: Sham technique in tibialis posterior

INTERVENTIONS:
Procedure: Deep dry needling in tibialis posterior — The inspector, with gloves, disinfects the area to be treated with 70º alcohol. Once the alcohol is applied, the intervenor locates and takes the myofascial trigger point and places the needle with the guide tube resting on the skin of the patient. The inspector holds the guide tube between the index and middle fingers lightly touch the needle with the index finger of the other hand to insert the needle perpendicularly into the skin, directing it towards the inspector's thumb. Once the needle is inserted subcutaneously, the guide tube is removed. The controller deepens the needle to myofascial trigger point, and makes fast inputs and outputs into it. The rapid exit is made to the subcutaneous cellular tissue, outside the muscle, but not outside the skin. Next, hemostasis is performed in the area. Once this hemostasis is completed, the patient is incorporated and dressed.
  Arms: Deep dry needling in tibialis posterior
Procedure: Sham technique in tibialis posterior — The patient lies on the stretcher without the trousers. The interventor, with the guide tube, simulates the technique of puncture in the right twin of the subject. The comptroller cleans the area with 70º alcohol. Once the alcohol is applied, he performs the simulated dry needling technique in a plane with his index and middle fingers with the guide tube. It is important that the subject has his head stuck in the hollow of the head of the stretcher throughout the technique to make a correct masking.
  Arms: Sham technique in tibialis posterior

SUMMARY:
This study aims to analyze the changes in plantar support after the technique of deep dry puncture in the posterior tibial. The data will be analyzed by a baropodometer which will record the possible changes in the footprint. The investigator will perform a pre-intervention measurement and 3 post-intervention measurements (immediately after the intervention, at 24 hours and at 72 hours)

ELIGIBILITY:
Inclusion Criteria:

* presence of myofascial trigger point in the posterior tibialis
* Accept participation in the study (signature of informed consent)
* Do not present any exclusion criteria

Exclusion Criteria:

* Do not present myofascial trigger point in the tibialis posterior.
* Suffering and / or having suffered from lower limb pathologies, deformities or orthopedic injuries that could alter the static and biomechanics.
* Not clearly identify the Myofascial trigger point in the tibialis posterior.
* Have been diagnosed with fibromyalgia, myelopathy or radiculopathy.
* Having contraindicated the technique of dry needling for suffering, for example, coagulation problems.
* Be pregnant.
* Have used analgesics 24 hours before participating in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2018-12-11 (Actual)

PRIMARY OUTCOMES:
Pain pressure threshold | 72 hours
  Amount of pressure (Kg/cm2) applied at the tibialis posterior myofascial trigger point site that elicit pain for the patient will be reported

SECONDARY OUTCOMES:
baropodometric measurements: footprint | 72 hours
  The investigator will be collected maximum pressure point in the footprint (g / cm)
baropodometric measurements: Average footprint pressure | 72 hours
  The investigator will be collected the average footprint pressure (g/cm)
baropodometric measurements: forefoot area | 72 hours
  The investigator will be collected the forefoot area (cm)
baropodometric measurements:forefoot load | 72 hours
  The investigator will be collected the forefoot load (%)
baropodometric measurements: forefoot pressure variation | 72 hours
  The investigator will be collected the forefoot pressure variation (%)
baropodometric measurements: rearfoot support surface | 72 hours
  The investigator will be collected the rearfoot support surface (cm)
baropodometric measurements: hindfoot load | 72 hours
  The investigator will be collected the hindfoot load ( %)
baropodometric measurements: areas of maximum pressure between the foot lines | 72 hours
  The investigator will be collected the areas of maximum pressure between the foot lines (g/cm)

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad CEU Cardenal Herrera, Valencia, Moncada, Spain

REFERENCES:
- See also: The University CEU-Cardenal Herrera is th first private university in the Valencian Community. It belongs to the Foundation San Pablo - CEU and is the leading educational organization in Spain with three Universities all over Spain — http://www.uchceu.es

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2013-03-18): https://cdn.clinicaltrials.gov/large-docs/28/NCT03756428/Prot_SAP_ICF_000.pdf